CLINICAL TRIAL: NCT02208557
Title: PREBIOUS Trial : A Multicenter Randomized Controlled Trial of Preventive Midline Laparotomy Closure With a Bioabsorbable Mesh for the Prevention of Incisional Hernia.
Brief Title: Usefulness of a Prothetic Absorbable Mesh in Incisional Hernia Prevention After Midline Laparotomy
Acronym: PREBIOUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PR(AG)220/2013
Record Dates: First submitted 2014-05-02; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Incisional Hernia
Keywords: Incisional hernia; prevention; laparotomy closure; absorbable mesh
MeSH Terms: conditions — Incisional Hernia | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Laparotomy closure will be done by continuous PDS suture following a SL:WL ratio of 4:1 only is used for midline laparotomy closure.
  Interventions: Radiation: Control CT; Other: Clinical Follow Up
- Reinforcement with Absorbable Mesh (Experimental): Closure of the midline laparotomy incision is reinforced with insertion of a rectangular segment (1 cm wide and the length corresponding to the incision) of a prosthetic commercially available GORE® BIO-A® Tissue Reinforcement prosthesis (W. L. Gore & Associates, Flagstaff, Arizona, USA) mesh. The BIO-A® prosthesis is inserted using a "sandwich" method between the edges of the incision and maintained in situ with a continuous polydioxanone (PDS) suture following a suture length to wound length (SL:WL) ratio of 4:1.
  Interventions: Procedure: Reinforcement with Absorbable Mesh; Radiation: Control CT; Other: Clinical Follow Up

INTERVENTIONS:
Procedure: Reinforcement with Absorbable Mesh
  Other Names: GORE® BIO-A® Tissue Reinforcement prosthesis; (W. L. Gore & Associates, Flagstaff, Arizona, USA) mesh.; LNE/G-MED (CE) 0459
  Arms: Reinforcement with Absorbable Mesh
Radiation: Control CT — At the end of the follow up (6 Months) a CT scan will be done. Radiologically the incisional hernia is defined as a solution of continuity of the linea alba seen on the abdominal CT scan with the patient at rest.
  The radiologist is blinded to the patient's history and the technique used for midline fascial closure.
Other: Clinical Follow Up — The presence of incisional hernia was evaluated by physical examination at scheduled clinical visits (3 and 6 months after surgery) Clinically, an incisional hernia is defined as the presence of a reducible bulge or protrusion at the laparotomy incision scar, palpable during the Valsalva maneuver.

SUMMARY:
Background: Development of an incisional hernia is one of the most frequent complications of midline laparotomies requiring reoperation. This paper presents the rationale, design, and study protocol for a randomized controlled trial, the aim of which was to evaluate the efficacy and safety of prophylactically placing a bioabsorbable synthetic mesh for reinforcement of a midline fascial closure.

Methods: The PREBIOUS trial (PREventive midline laparotomy closure with a BIOabsorbable mesh) is a multicenter randomized controlled trial in which adult patients undergoing elective or urgent open abdominal operations through a midline laparotomy incision are assigned to one of two groups based on the laparotomy closure procedure: an intervention group in which a continuous polydioxanone (PDS) suture is reinforced with a commercially available GORE® BIO-A® Tissue Reinforcement prosthesis (W. L. Gore & Associates, Flagstaff, Arizona, USA), or a control group with continuous PDS suture only. Both groups are followed over 6 months.

Outcomes: The primary outcome is the appearance of incisional hernias assessed by physical examination at clinical visits and radiologically (CT scan) performed at the end of follow-up. Secondary outcomes are the rate of complications, mainly infection, hematoma, burst abdomen, pain, and reoperation. The PREBIOUS trial has the potential to demonstrate that suture plus prosthetic mesh insertion for routine midline laparotomy closure is effective in preventing incisional hernias after open abdominal surgery, to avoid the effects on those affected, such as poor cosmesis, social embarrassment, or impaired quality of life, and to save costs potentially associated with incisional hernia surgical repair.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older,
* Signed informed consent,
* Patients undergoing elective or urgent open abdominal surgical procedures regardless of benign or malignant disease.

Exclusion Criteria:

* Presence of primary or recurrent incisional hernia
* Expected survival < 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of incisional hernia | 6 months
  The primary endpoint is the incidence of incisional hernia, either symptomatic or asymptomatic in the mesh and suture-only groups. Because appearance of an incisional hernia occurs within the first months after laparotomy, assessment of efficacy was carried out during scheduled clinical visits over a period of 6 months. The presence of incisional hernia was evaluated by physical examination at scheduled clinical visits and radiologically by an abdominal CT scan performed at the end of follow-up (6 months after operation).

SECONDARY OUTCOMES:
Perioperative complications | 30 days
  Secondary endpoints are perioperative complications, including wound infection, hematoma, eventration, pain, reoperation.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Lopez-Cano, MD, PhD, Principal Investigator — Hospital Universitari Vall d´Hebrón
Locations (6):
- Spain (6):
  - Hospital del Mar, Parc de Salut Mar, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital de Igualada, Igualada, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital Arnau de Vilanova, Lleida, Lerida
  - Hospital de Sagunto, Sagunto, Valencia